CLINICAL TRIAL: NCT06667336
Title: The Impact of Suctioning on Oxygenation During RSI in the Emergency Department-A Multi-Center Pilot Study
Brief Title: The Impact of Suctioning on Oxygenation During RSI in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-01-32
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: RSI
Keywords: RSI; Emergency Department; Resuscitation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Suction (Active Comparator): This suction was applied only as needed to clear secretions
  Interventions: Procedure: intermittent suction
- Continuous Suction (Active Comparator): The suction catheter was inserted at the start of laryngoscopy and maintained in the oropharynx until the moment of ETT delivery
  Interventions: Procedure: continuous suction

INTERVENTIONS:
Procedure: intermittent suction — This suction was applied only as needed to clear secretions
  Arms: Intermittent Suction
Procedure: continuous suction — The suction catheter was inserted at the start of laryngoscopy and maintained in the oropharynx until the moment of ETT delivery.
  Arms: Continuous Suction

SUMMARY:
Rapid Sequence Intubation (RSI) is a common procedure in Emergency Departments (ED). However, it is a high-risk procedure and has been associated with significant complications including hypoxia, hypotension, airway trauma, aspiration, and death. Specifically, hypoxic episodes during intubation can lead to poor outcomes such as dysrhythmias, haemodynamic compromise, hypoxic brain injury and cardiac arrest, and is therefore of primary concern during any intubation procedure. Aspiration is a serious adverse event and potential cause of hypoxia during RSI and can lead to poor patient outcomes downstream of the procedure. The reported incidence of aspiration during RSI in the ED ranges from 3 to 8% in the ED population. In order to achieve an optimal view of the glottis and prevent pulmonary aspiration of fluids in the oropharynx, providers apply suction prior to and during laryngoscopy, using a Yankauer or large-bore suction catheter.

There is currently significant variation in suctioning during laryngoscopy, with some providers using very little suction as needed to clear heavy fluids (judicious suctioning), while others utilise suction aggressively (lead with suction) and as a part of their routine laryngoscopy technique. Evidence suggests inline suction on already-intubated patients accelerates desaturation, but we are aware of no studies examining the impact suctioning has on the speed of desaturation during emergent endotracheal intubation.

This pilot study aims to compare the effects of intermittent, as-needed "judicious" suctioning versus aggressive "continuous" (lead with) suctioning on oxygenation during rapid sequence intubation in the emergency department.

DETAILED DESCRIPTION:
Intervention

The aim of this study is to investigate the effect of suctioning (a current technique used conventionally in RSI) on oxygenation levels during RSI. This being noted, there is no new intervention being applied to the patient.

In order to investigate this, the current standard of care of suctioning will be used either by judicious means (i.e. in and out suction as needed) or continuous means (i.e. throughout the procedure, including laryngoscopy and tube placement) according to conventional practice at the discretion of the treating physician. For all patients involved in the study, there will be no new intervention applied. The impact of the use of suctioning, again which is standard of care and applied by convention, will be determined by measuring oxygen saturation as a primary outcome. All aspects of RSI will be at the discretion of the treating clinician, which is the current standard, including induction/relaxant medication, positioning of the patient, preoxygenation method, method of intubation and post-intubation sedation. At all institutions RSI is performed in a similar manner utilising an airway checklist (Appendix 1 and 2). However, there are no 'Standard Operating Procedures' for RSI in any ED and therefore intubation technique will vary depending on clinician preference and the clinical circumstances.

Once the decision to perform RSI has been made by the treating team, the patient will be enrolled into either a judicious or continuous suction group at random. In either case, suctioning will be applied to the patient as determined necessary by the clinician. Rapid sequence intubation will then be performed in the standard means by the treating provider.

Data Collection

The data will be collected prospectively during the time of RSI by nursing and medical staff with the use of a data collection sheet. Staff at RPA ED are familiar with the data collection sheets as prior studies in relation to RSI have been performed previously (Study number Re: X12- 0394). Similarly, staff at Lincoln Medical Center and Mount Sinai perform routine data collection on all RSI's performed in the ED for quality improvement purposes.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine Patients
* Requiring Rapid Sequence Intubation in the Resuscitation Bay
* 18 years+

Exclusion Criteria:

* Patients that have a heavily soiled airway (i.e. secretions, vomitus, blood)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation achieved (SpO2) | 10 minutes
  the oxygen saturation achieved (SpO2) at the time of tube placement (via confirmation with first ETCO2 waveform) achieved during the intubation period.

SECONDARY OUTCOMES:
Incidence of Desaturation | 2 minutes
  Incidence of desaturation (SaO2 <90%) or >10 points from baseline during the intubation period
Lowest O2 Saturation | 2 minutes
  Lowest O2 saturations at any point during the intubation period
End-Tidal Oxygen Concentration ( ETO2) | 2 minutes
  The ETO2 at induction and at Endotracheal Tube (ETT) confirmation.
Time from Preoxygenation | 5 minutes
  Time from preoxygenation to endotracheal intubation
Complications During RSI | 1 minute
  Complications during RSI: bradycardia, tachycardia, hypotension, hypertension, oesophageal intubation, aspiration, airway or dental trauma, equipment or medication error
Intubation Attempts | 1 minute
  Number of intubation attempts

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT06667336/Prot_SAP_000.pdf